CLINICAL TRIAL: NCT04480814
Title: A Clinical Performance Study to Validate the Use of Novel Molecular Diagnostic Assays for the Detection of Cancer Biomarkers in Peripheral Blood and Primary Tumor Tissue Samples of Patients With Metastatic ER+/HER2- Breast Cancer
Brief Title: Validation of Molecular Diagnostic Assays to Detect Cancer Biomarkers in Blood & Primary Tumor in ER+/HER2- MBC
Status: Completed | Type: Observational
Sponsor: Pharmassist Ltd (Industry)
Collaborators: University of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: CBS-PIK3CA
Record Dates: First submitted 2020-02-20; First posted 2020-07-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Liquid biopsy; CTC; Plasma; PIK3CA
MeSH Terms: conditions — Breast Neoplasms; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CTCs, plasma-ctDNA and primary tumor tissue samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metastatic Breast Cancer: The study population are subjects with a confirmed diagnosis of ER+/HER2 metastatic Breast Cancer patient before the treatment initiation.
  The selected inclusion/exclusion criteria have been set to include in the performance study appropriate population of interest, as broad as possible, but to exclude these subjects that have another current malignancy or any history of recent malignancy within 3 years.
  Interventions: Diagnostic Test: PIK3CA kit
- Healthy volunteers: In case of healthy volunteers only peripheral blood samples will be collected.
  Interventions: Diagnostic Test: PIK3CA kit

INTERVENTIONS:
Diagnostic Test: PIK3CA kit — Prospective investigation of clinical samples for evaluation of IVD clinical performance

SUMMARY:
Conventional biopsy and surgical tumor resection are invasive procedures that capture only one instance of the progression of the tumor. However, the genome of tumor is not static, but it is constantly altered during treatment.

Liquid biopsy is a non-invasive approach based on the extraction of information through peripheral blood analysis. It makes it possible to characterize the development of a solid tumor in real time, through detailed molecular analysis of circulating genetic material in peripheral blood.

DETAILED DESCRIPTION:
Conventional biopsy and surgical tumor resection are invasive procedures that capture only one instance of the progression of the tumor. However, the genome of tumor is not static, but it is constantly altered during treatment.

Liquid biopsy is a non-invasive approach based on the extraction of information through peripheral blood analysis. It makes it possible to characterize the development of a solid tumor in real time, through detailed molecular analysis of circulating genetic material in peripheral blood.

Study procedure:

1. Initial Visit (V0-Baseline): For the purposes of the study the following information will be collected: the demographics, medical and social history, the characteristics of the disease (stage, molecular characterization e.t.c) and the treatment regimen that is followed. As part of the visit, 20 mL of peripheral blood will be drawn prior to their treatment according to physician's suggestion as per common clinical practice. Blood samples will be then sent to ACTC laboratory for plasma/CTC isolation, DNA and RNA extraction and subsequent test for biomarkers. Primary tumor tissue samples will be also collected
2. Follow-up visit (V1): Response to treatment by RECIST based on restaging CTs/MRIs will be documented during this visit, which will take place 3 months after treatment initiation. As part of the visit, 20 mL of peripheral blood will be drawn.

Blood samples will be then sent to laboratory for plasma/CTC isolation, DNA and RNA extraction and subsequent test for biomarkers. Survival status and clinical response (CR, PR, SD, PD) will be also documented.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥ 18 years of age.
2. Histological confirmed ER+/HER2- metastatic Breast Cancer prior to beginning a treatment
3. Life expectancy permits participation to the study.
4. Available tumor tissue sample for molecular analysis.
5. Signed informed consent form.

Exclusion Criteria:

1. Female younger than 18 years old.
2. History of another malignancy within 3 years or current 2nd primary malignancy.
3. Patients that have not signed the informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 120 with metastatic breast cancer 30 healthy subjects
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Clinical performance of PIK3CA kit in CTCs, plasma and tumor tissue samples of metastatic breast cancer patients | 18 months
  The performance of PIK3CA kit on detecting mutations in CTCs samples of metastatic breast cancer patients will be assessed via Sensitivity, Specificity, Positive and Negative Predictive Values, Positive and Negative Likelihood Ratios, Accuracy and Diagnostic Odds Ratio. The point of primary evaluation in CTCs samples will be at baseline and droplet digital PCR will be used as reference method.
  The performance of PIK3CA kit on detecting mutations in plasma-ctDNA, and tumor tissue samples of metastatic breast cancer patients will be assessed via Sensitivity, Specificity Positive and Negative Predictive Values, Positive and Negative Likelihood Ratios, Accuracy and Diagnostic Odds Ratio. The point of primary evaluation in plasma-ctDNA and tumor tissue samples will be at baseline and therascreen PIK3CA RGQ PCR Kit will be used as reference method.

SECONDARY OUTCOMES:
- To study the PIK3CA Mutation Status before and after treatment of metastatic breast cancer patients using PIK3CA kit. | 24 months
  Presence of PIK3CA mutations at a second visit following to baseline of metastatic breast cancer patients using the PIK3CA kit.
- To assess the PIK3CA Mutation Status before treatment vs treatment response of metastatic breast cancer patients using PIK3CA kit. | 24 months
  Association of PIK3CA mutations presence at baseline with clinical response to treatment (CR, PR, SD, PD) of metastatic breast cancer patients using PIK3CA kit.
- To correlate patients' survival status with PIK3CA mutations at baseline | 24 months
  Metastatic breast cancer patients' survival status by presence of PIK3CA mutations at baseline.

OTHER OUTCOMES:
To study CK-19 expression in CTC samples | 24 months
  Detection of CK-19 expression in CTCs
To study methylation status of ESR1 in CTC, ctDNA and tumor tissue samples | 24 months
  Methylation status of ESR1 in CTC, plasma and tumor samples
To study the presence of other biomarkers in tissue and liquid biopsy sample (at baseline). | 24 months
  Molecular profile of cancer biomarkers between tissue and peripheral blood samples

CONTACTS AND LOCATIONS:
Locations (4):
- Greece (4):
  - University General Hospital of Alexandroupoli, Alexandroupoli, Alexandroupolis
  - Aretaieio University Hospital of Athens, Athens, Attica
  - University General Hospital of Athens Attikon, Athens, Attica
  - Metropolital Hospital, Piraeus, Piraeus